CLINICAL TRIAL: NCT03883126
Title: Remote Alcohol Monitoring to Facilitate Abstinence Reinforcement With an Underserved Population
Brief Title: Remote Alcohol Monitoring to Facilitate Abstinence From Alcohol: Exp 1
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mikhail N Koffarnus (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Mikhail N Koffarnus, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 54073; R01AA026605 (NIH)
Record Dates: First submitted 2019-03-15; First posted 2019-03-20 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group A (Active Comparator): Group A will receive nearly immediate monetary payments over the internet each day they remotely provide negative breathalyzer samples, but will not receive the payments if they provide positive samples or fail to provide samples in a timely manner for the first 3 weeks of the intervention. For the remaining 9 weeks they will continue to receive incentives for submitting negative samples.
  Interventions: Behavioral: Contingency management
- Group B (Active Comparator): Group B will receive nearly immediate monetary payments over the internet each day they remotely provide negative breathalyzer samples, but will not receive the payments if they provide positive samples or fail to provide samples in a timely manner for the first 3 weeks of the intervention.For the remaining 9 weeks they will not be required to submit breathalyzer samples.
  Interventions: Behavioral: Contingency management
- Group C (Sham Comparator): Group C will receive nearly immediate monetary payments over the internet each day they remotely provide breathalyzer samples regardless of the alcohol content, but will not receive the payments if they fail to provide samples in a timely manner for the first 3 weeks of the intervention. For the remaining 9 weeks they will continue to receive incentives for submitting on time samples regardless of alcohol content.
  Interventions: Behavioral: Contingency management
- Group D (Sham Comparator): Group D will receive nearly immediate monetary payments over the internet each day they remotely provide breathalyzer samples regardless of the alcohol content, but will not receive the payments if they fail to provide samples in a timely manner for the first 3 weeks of the intervention. For the remaining 9 weeks they will not be required to submit breathalyzer samples.
  Interventions: Behavioral: Contingency management
- Group E (No Intervention): Group E will have no intervention, they will only complete assessment sessions.

INTERVENTIONS:
Behavioral: Contingency management — Monetary incentives are delivered to participants contingent upon on-time breathalyzer submissions and verified abstinence from alcohol.
  Other Names: Contingent incentives
  Arms: Group A; Group B
Behavioral: Contingency management — Monetary incentives are delivered to participants contingent upon on-time breathalyzer submissions only with no contingency on alcohol use.
  Other Names: Noncontingent incentives
  Arms: Group C; Group D

SUMMARY:
Directly reinforcing abstinence from alcohol with monetary incentives is an effective treatment for alcohol dependence, but barriers in obtaining frequent, verified biochemical measures of abstinence limit the dissemination of this treatment approach. The goal of this study is to use technological advancements to remotely, accurately, and securely monitor alcohol use with a newly developed smartphone app and breathalyzer. This treatment approach has the potential to facilitate the dissemination of an effective, evidence-based treatment for alcohol dependence to a broader population whose treatment needs are not currently being adequately met.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual (DSM)-5 criteria for alcohol use disorder
* Average 3 or more heavy drinking days (≥5 drinks in one occasion for men, ≥4 for women) per week for the past month on the Timeline Follow-back.
* Must endorse alcohol as their primary drug of use.
* Express a desire to abstain from drinking.

Exclusion Criteria:

* Are currently enrolled in an alcohol treatment program (not including attendance at Alcoholics Anonymous or similar community support meetings).
* Score 23 or greater on the Alcohol Withdrawal Symptom Checklist, a score indicating that medication would be likely required to manage alcohol detoxification.
* Pregnant women, lactating women, or women who are planning to become pregnant in the next 15 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Pattern of abstinence from alcohol during intervention | up to 66 weeks
  Breathalyzer assessments will be collected during the treatment period. This outcome measure will consist of the percentage of days without alcohol use as detected by the breathalyzers.
Treatment acceptability | A total of 12 assessment sessions spanning over a 66 week period.
  Participant ratings of treatment acceptability on a customized questionnaire will be collected during assessment sessions

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Nationwide Online Enrollment from the Unversity of Kentucky, Lexington, Kentucky
  - University of Kentucky Turfland: In-person enrollment, Lexington, Kentucky
  - Carilion Clinic: In person-enrollment, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Final research data for this project will be made as available as possible, while safeguarding the privacy of participants and protecting all confidential and proprietary data. Data will be available for use after the main findings from the final dataset have been accepted for publication. The data and associated documentation will only be made available to users under a Data Use Agreement that provides for 1) a commitment to using the data only for research purposes and not to identify any individual participant and 2) a commitment to destroying or returning the data after analyses are completed. To ensure compliance with HIPAA regulations, only a Limited Data Set will be available for use. The method of data release will be determined on a case-by-case basis depending upon the amount and type of data required.
Supporting Information: Study Protocol, SAP, ICF